CLINICAL TRIAL: NCT06226285
Title: Quality of Life for Carers Through a Person-Centred Technological Solution
Acronym: TechQoL4Carers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade da Coruña (Other)
Collaborators: Ministry of Science and Innovation, Spain (Other Government); Center on Information and Communication Technologies (Other)
Responsible Party: Principal Investigator, Betania Groba González, Associate Professor in Occupational Therapy-Nursing, PhD in Health Sciences, Universidade da Coruña
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2023_019
Record Dates: First submitted 2024-01-03; First posted 2024-01-26 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Informal Caregivers; Quality of Life; Technology; Activities of Daily Living
Keywords: Quality of Life; informal caregivers; innovation; technological solution; wearable devices; occupational balance; self-management of health; empowerment; person-centred care; participatory processes
MeSH Terms: conditions — Empowerment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Informal caregivers (Experimental): Informal caregivers will participate in a participatory process of development, testing and validation of a technological platform aimed at improving their quality of life, impact of care, occupational balance, self-management of health and empowerment.
  Interventions: Device: TechQoL4Carers Platform

INTERVENTIONS:
Device: TechQoL4Carers Platform — The TechQoL4Carers platform is a technological solution that has been designed and developed by the research team in collaboration with the end users. A website and a mobile application integrate the platform. The services offered are: summary of the person's state of health; training content, advice and personalised recommendations based on their situation in terms of quality of life, provision of care, occupational balance, self-management of health and empowerment. It also allows synchronisation with the Xiaomi Smart Band 7/8 activity wristband.
  The intervention has a duration of three months. Participants will use the services of TechQoL4Carers and wear the Xiaomi Smart Band 7/8 wristband on a regular basis.
  It is expected that caregivers will access and use the TechQoL4Carers platform, at least once a week, to answer the weekly questionnaire and they will consult, at least once a month, the training contents for self-care and for the provision of care.

SUMMARY:
This study is entitled Quality of Life for Carers through a Person-Centred Technological Solution, whose acronym is TechQoL4Carers.

The goal of this pilot study is to develop an innovative technological solution (TechQoL4Carers) to improve the Quality of Life (QoL), occupational balance, impact of care, self-management of health, and empowerment of informal caregivers of older people or people with disability. The main question it aims to answer is: Will the routine use of TechQoL4Carers platform have a positive impact on the daily life of informal caregivers? The study will examine these variables in a specific way: QoL, impact of care and burden, occupational balance, health self-management, and empowerment.

Informal caregivers will participate in a participatory process of development, testing and validation of the technological platform TechQoL4Carers. At the beginning and end of the study, participants will be asked to answer questionnaires to capture their perspective on the central variables of the study and on the utility and usability of the technology. Then, for three months, participants will:

* use TechQoL4Carers platform on their mobile phone or computer,
* wear the Xiaomi Smart Band 7/8,
* provide weekly reports of health and care related quality of life,
* and receive personalized recommendations and training materials.

At the end, they will also participate in an in-depth interview on the impact of the project on their daily activities.

DETAILED DESCRIPTION:
The project was submitted to the 2021 Call for Strategic Projects oriented to the Ecological and Digital Transition of the Spanish Ministry of Science and Innovation, of the State Plan for Scientific, Technical and Innovation Research 2021-2023, which, in turn, is part of the National Recovery, Transformation and Resilience Plan, with funding from Next Generation funds of the European Union.

The technological solution will offer training contents for informal caregivers, which will enable them to increase their knowledge and acquire new skills, including digital ones, so that this proposal will also contribute to the promotion of education, lifelong learning and skills development. In this way, the TechQoL4Carers project will break the digital divide and promote digital inclusion, through an inclusive and sustainable service that put people at the centre.

The social challenge to which the project responds is the QoL of caregivers. In Spain, 15.3% of the population is in an informal caregiver role. The latest data from 2020 show that 53% of Spanish informal caregivers spend 20 hours or more per week caring, represented by women (58%) and aged between 45 and 64 years (52%). The impact of informal care on people's everyday life is double sided: on the one hand, there is evidence of positive aspects, but on the other hand, negative aspects are reflected on different levels (mental, physical, economic and social). This situation has aggravated due to the global COVID-19 pandemic. Nowadays, health, social and care systems for informal caregivers are needed from a person-centred perspective to promote their health, QoL and empowerment. Technology is a promising tool to provide personalised services for active participation in these processes.

TechQoL4Carers is based on a person-centred development, participatory design techniques and an iterative procedure to obtain the final version of the platform. This platform will consist of a website, interconnected with a mobile application and wearable devices, which will offer a set of personalised services that will allow end users to collect and monitor data on their own QoL, occupational balance and healthy lifestyle; to receive personalised warnings; and to access e-training content as additional support in their care tasks and in their own self-care.

It is structured in 7 Work Packages (WP), aligned with the objectives and developed in specific tasks and deliverables. Three main research stages are highlighted: analysis of evidence and definition of requirements (WP1 and WP2); development of the platform and its integration with wearable devices, artificial intelligence and cybersecurity (WP3 and WP4); and validation of the platform and knowledge generation (WP5 and WP6). For the design, testing and validation of the platform (WP5) a pilot study will be conducted following a mixed methodology (quantitative and qualitative). Questionnaires and interviews as well as testing of the platform will be conducted with informal caregivers in order to obtain a final product that considers the end-user in the whole process.

These results are expected to have a scientific and social impact. Knowledge and evidence will be generated on how to improve the QoL of informal caregivers through technology, providing them with tools that will enable more efficient time management and occupational balance. This can indirectly improve the QoL and wellbeing of the people receiving their care (mainly, older people or people with disability).

ELIGIBILITY:
Inclusion Criteria:

* Be 18 years of age or older.
* Perform the role of informal caregiver, being the main caregiver.
* To be living with the person receiving the care.
* Regularly use a smartphone.
* Commit to using the activity wristband on a regular basis during the project development period.

Exclusion Criteria:

* Have been an informal caregiver for less than one year.
* Be the main caregiver of more than one person in a situation of dependency.
* Have modified legal capacity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2025-03-24 (Actual)

PRIMARY OUTCOMES:
Change in health-related Quality of Life from baseline to post-intervention | Pre-Post: baseline and one-month post-intervention
  Health-related Quality of Life (QoL) will be measured through the self-administered tool EuroQol 5 dimensions 5 levels (EQ-5D-5L).
  Health state is obtained from the EQ-5D-5L, through its descriptive system with five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. The dimensions are scored on a 5-point Likert scale reflecting the level of severity (no problem, slight problems, moderate problems, severe problems, and extreme problems or unable to perform). The health profile or health state describes the level of severity that the person perceives in each dimension and it is represented through an individual code for each dimension scored between 1 and 5 or through a single five-digit code (ranging from 11111 to 55555).
Change in overall health from baseline to post-intervention | Pre-Post: baseline and one-month post-intervention
  Health-related QoL will be measured through the self-administered tool EQ-5D-5L.
  Overall health is derived from a visual analogue scale (VAS) on perceived health, from 0 to 100. In this way, the person scores his or her health on a given day; assigning it a value between 0 (the worst health you can imagine) and 100 (the best health you can imagine).
Change in care-related QoL from baseline to post-intervention | Pre-Post: baseline and one-month post-intervention
  Care-related QoL will be measured through the dimensions of the Care-related QoL instrument (CarerQol).
  The seven dimensions (CarerQol-7D) are fulfillment, relational, mental health, social, financial, perceived support, and physical dimension. They are scored on a Likert scale with three values (1 to 3) indicating the level of severity (no, some, and a lot). Score range: 7 to 21. Score interpretation: The higher the score on the dimensions, the worse the impact of care on the life of the caregiver.
Change in perceived well-being from baseline to post-intervention | Pre-Post: baseline and one-month post-intervention
  Well-being related to care-related QoL will be measured through the visual analogue scale (VAS) of the Care-related QoL instrument (CarerQol).
  The CarerQol-VAS allows rating how happy the person feels at that moment as a measure of general well-being. This construct is scored on a range from 0 (completely unhappy) to 10 (completely happy). Score interpretation: The higher the score, the better the situation in terms of the impact of care.

SECONDARY OUTCOMES:
Change in caregiver burden from baseline to post-intervention | Pre-Post: baseline and one-month post-intervention
  The Zarit Burden Interview (ZBI) is a questionnaire designed for the caregiving population to assess the level of burden and to detect possible caregiving stressors. The 22-item version is used, scored from 1 to 5. Score range: 22 to 110. Score interpretation with two cut-off points: no burden, 22 to 46 points; mild burden, 47 to 55 points; and severe burden, 56 to 110 points.
Change in caregiver strain from baseline to post-intervention | Pre-Post: baseline and one-month post-intervention
  The Caregiver Strain Index (CBI) or Robinson Index is a 13-item tool for caregivers to measure perceived strain, and detect burden and possible stressors related to caregiving. Each item is answered in a dichotomous way: yes or no. Score range: 0 to 13. Score interpretation: Scores of 7 or more, identify caregivers at risk for high caregiving strain or burden.
Change in occupational balance from baseline to post-intervention | Pre-Post: baseline and one-month post-intervention
  Occupational balance will be measured through the Occupational Balance Questionnaire, Spanish version (OBQ-E).
  This self-administered tool of 13 items is scored on a six-step ordinal scale, ranging from 0 (completely disagree) to 5 (completely agree). It evaluates the person's current experience with occupational balance. Score range: 0 to 65. Score interpretation: The results show that the higher the score, the higher the occupational balance.
Change in perceived empowerment from baseline to post-intervention | Pre-Post: baseline and one-month post-intervention
  The Psychological Empowerment Instrument (PEI) will be used to assess changes in informal caregivers' perceptions of empowerment.
  It is a self-administered instrument that measures psychological empowerment in the work environment, considering four cognitive dimensions: competence, meaning, self-determination, and impact. The Spanish version of the PEI comprises 13 items divided among the four dimensions and scored on a 7-point Likert scale. This version will be used in the study replacing the references to work and the role of the workers with terms associated with care and caregivers. Score range: 7 to 91 points. Score interpretation: The higher the score, the higher the level of psychological empowerment.
Change in physical activity measured by the Xiaomi Smart Band during intervention | 3 months wearing the Xiaomi Smart Band
  In the study, participants will use the Xiaomi Smart Band activity wristband regularly during the three months of the intervention. Versions 7 and 8 of the Xiaomi Smart Band activity wristband allow the recording and monitoring of health-related variables: physical activity, sleep, heart rate, blood oxygen saturation (SpO₂), women's health, and stress.
  The wristband will be synchronized with the TechQoL4Carers platform to monitor physical activity: number of steps, distance in meters, and activity in minutes.
Change in sleep measured by the Xiaomi Smart Band during intervention | 3 months wearing the Xiaomi Smart Band
  In the study, participants will use the Xiaomi Smart Band activity wristband regularly during the three months of the intervention. Versions 7 and 8 of the Xiaomi Smart Band activity wristband allow the recording and monitoring of health-related variables: physical activity, sleep, heart rate, blood oxygen saturation (SpO₂), women's health, and stress.
  The wristband will be synchronized with the TechQoL4Carers platform to monitor sleep: light sleep, deep sleep, REM sleep, and time awake after sleep onset in minutes.
Change in daily functioning measured by TechQoL4Carers platform during the intervention | Once a week during the intervention (three months)
  The TechQoL4Carers platform allows the self-administration of a weekly questionnaire designed by the research team to identify changes perceived by the person in daily functioning based on the variables studied: quality of life, satisfaction with the care, occupational balance, self-management of health, and empowerment.
  The development of this questionnaire has been based on previous surveys developed by the research team, but it has been adapted to caregivers for this study.
  The TechQoL4Carers weekly questionnaire is integrated with nine items that are answered using a six-point Likert scale, ranging from 0 (completely disagree) to 5 (completely agree). Score range: 0 to 45 points. Score interpretation: The higher the score, the greater the perception of positive changes in quality of life-related factors.
TechQoL4Carers Satisfaction Questionnaire | One month post-intervention
  The TechQoL4Carers Satisfaction Questionnaire will be administered at the end of the intervention to assess end-user satisfaction with the project and the technology. The questionnaire has been adapted for this study based on the Technology Satisfaction Factor Loadings questionnaire (Njoroge et al., 2012).
  It is a self-administered questionnaire consisting of 16 items grouped into four factors (proficiency, assessment, performance, and TechQoL4Carers platform), rated on a six-point scale, ranging from 0 (completely disagree) to 5 (completely agree). Score range: 0 to 80. Score interpretation: The higher the agreement with the statements, the higher the satisfaction with the project.
Meaning attributed to participation in the project | One month post-intervention
  At the end of the project, a semi-structured individual interview will be conducted with each caregiver. The interview guide has been designed to elicit the meaning that the caregivers give to the caregiving experience, to the participation in the project, to the use of technology in the project, and the impact of this project on their daily life (quality of life, impact of caregiving, occupational balance, self-management of health and empowerment).
  This interview will take place in the collaborating entities, in a quiet and comfortable place, and at a time that suits the needs of the participants. It will be recorded with a digital device to facilitate the literal transcription. This information will be coded and at the end of the study, the transcriptions will be anonymized and the audios will be deleted.

CONTACTS AND LOCATIONS:
Overall Officials: Betania Groba, PhD, Principal Investigator — Universidade da Coruña; Laura Nieto-Riveiro, PhD, Principal Investigator — Universidade da Coruña; Javier Pereira, PhD, Study Chair — Universidade da Coruña
Locations (1):
- Universidade da Coruña, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be available for sharing with the scientific community, upon request and after the acceptance for publication of the main findings from de final data set.
  The data will be completely anonymized for sharing. The dataset will include only the results of quantitative variables. An institutional data use agreement will be required before data is shared.
  The microdata will also be transferred to the specific Social Studies Data Bank of the Spanish Sociological Research Center.
Supporting Information: Study Protocol
Time Frame: The data will be available after the acceptance for publication of the main findings from de final data set. Time frame estimated: June 2025.
Access Criteria: Data will be available upon request to the principal investigators. Requests should be emailed to: b.groba@udc.es and laura.nieto@udc.es

REFERENCES:
- [Background] Bretones FD, Jáimez MJ. Spanish adaptation and validation of the Psychological Empowerment Scale. Interdisciplinaria. 2022; 39(1): 195-210. https://doi.org/10.16888/INTERD.2022.39.1.12
- [Background] Brouwer WB, van Exel NJ, van Gorp B, Redekop WK. The CarerQol instrument: a new instrument to measure care-related quality of life of informal caregivers for use in economic evaluations. Qual Life Res. 2006 Aug;15(6):1005-21. doi: 10.1007/s11136-005-5994-6. PMID 16900281
- [Background] Concheiro-Moscoso P, Groba B, Martinez-Martinez FJ, Miranda-Duro MDC, Nieto-Riveiro L, Pousada T, Queiros C, Pereira J. Study for the Design of a Protocol to Assess the Impact of Stress in the Quality of Life of Workers. Int J Environ Res Public Health. 2021 Feb 3;18(4):1413. doi: 10.3390/ijerph18041413. PMID 33546392
- [Background] Concheiro-Moscoso P, Groba B, Martinez-Martinez FJ, Miranda-Duro MDC, Nieto-Riveiro L, Pousada T, Pereira J. Use of the Xiaomi Mi Band for sleep monitoring and its influence on the daily life of older people living in a nursing home. Digit Health. 2022 Aug 29;8:20552076221121162. doi: 10.1177/20552076221121162. eCollection 2022 Jan-Dec. PMID 36060611
- [Background] EuroQol Research Foundation. EQ-5D-5L User Guide Basic information on how to use the EQ-5D-5L instrument. 2019. https://euroqol.org/publications/user-guides/
- [Background] Hernandez G, Garin O, Pardo Y, Vilagut G, Pont A, Suarez M, Neira M, Rajmil L, Gorostiza I, Ramallo-Farina Y, Cabases J, Alonso J, Ferrer M. Validity of the EQ-5D-5L and reference norms for the Spanish population. Qual Life Res. 2018 Sep;27(9):2337-2348. doi: 10.1007/s11136-018-1877-5. Epub 2018 May 16. PMID 29767329
- [Background] López AS, Moral SM. Validación del Índice de Esfuerzo del Cuidador en la población española [Validation of the Caregiver Strain Index in Spanish population]. Enferm Comunitaria. 2005; 1(1): 12-17.
- [Background] Martín-Carrasco M, Salvadó I, Nadal Álava S, Miji LC, Rico JM, Lanz P, Taussig MI. Adaptación para nuestro medio de la escala de sobrecarga del cuidador (Caregiver Burden Interview) de Zarit. Revista de Gerontología. 1996; 6(4): 338-346.
- [Background] Martin-Carrasco M, Otermin P, Perez-Camo V, Pujol J, Aguera L, Martin MJ, Gobartt AL, Pons S, Balana M. EDUCA study: Psychometric properties of the Spanish version of the Zarit Caregiver Burden Scale. Aging Ment Health. 2010 Aug;14(6):705-11. doi: 10.1080/13607860903586094. PMID 20544413
- [Background] Miranda-Duro MDC, Nieto-Riveiro L, Concheiro-Moscoso P, Groba B, Pousada T, Canosa N, Pereira J. Analysis of Older Adults in Spanish Care Facilities, Risk of Falling and Daily Activity Using Xiaomi Mi Band 2. Sensors (Basel). 2021 May 11;21(10):3341. doi: 10.3390/s21103341. PMID 34064993
- [Background] Njoroge J, Norman A, Reed D, Suh I. Identifying Facets of Technology Satisfaction: Measure Development and Application. J Learn High Educ. 2012; 1(2): 7-17. https://eric.ed.gov/?id=EJ1145014
- [Background] Odriozola Gojenola M, Vita Garay A, Maiz Alkorta B, Zialtzeta Aduriz L, Bengoetxea Gallastegi L. Índice de esfuerzo del cuidador: test diagnóstico de sobrecarga en cuidadores de enfermos con demencia. Semer - Med Fam. 2008; 34(9): 435-438. https://doi.org/10.1016/S1138-3593(08)75201-8
- [Background] Peral-Gomez P, Lopez-Roig S, Pastor-Mira MA, Abad-Navarro E, Valera-Gran D, Hakansson C, Wagman P. Cultural Adaptation and Psychometric Properties of the Spanish Version of the Occupational Balance Questionnaire: An Instrument for Occupation-Based Research. Int J Environ Res Public Health. 2021 Jul 14;18(14):7506. doi: 10.3390/ijerph18147506. PMID 34299957
- [Background] Ramos-Goni JM, Craig BM, Oppe M, Ramallo-Farina Y, Pinto-Prades JL, Luo N, Rivero-Arias O. Handling Data Quality Issues to Estimate the Spanish EQ-5D-5L Value Set Using a Hybrid Interval Regression Approach. Value Health. 2018 May;21(5):596-604. doi: 10.1016/j.jval.2017.10.023. Epub 2017 Dec 2. PMID 29753358
- [Background] Robinson BC. Validation of a Caregiver Strain Index. J Gerontol. 1983 May;38(3):344-8. doi: 10.1093/geronj/38.3.344. PMID 6841931
- [Background] Spanish Ministry of Health. Spanish National Health Survey 2011/2012. 2012. https://www.sanidad.gob.es/estadEstudios/estadisticas/encuestaNacional/encuesta2011.htm
- [Background] Spreitzer GM. Psycological, Empowerment in the Workplace: Dimensions, Measurement and Validation. Acad Manag J. 1995; 38(5): 1442-1465. https://doi.org/10.2307/256865
- [Background] Spreitzer GM. Social structural characteristics of psychological empowerment. Acad Manag J. 1996; 39(2): 483-504. https://doi.org/10.2307/256789
- [Background] Wagman P, Hakansson C. Exploring occupational balance in adults in Sweden. Scand J Occup Ther. 2014 Nov;21(6):415-20. doi: 10.3109/11038128.2014.934917. Epub 2014 Aug 6. PMID 25100158
- [Background] Xiaomi. Xiaomi Smart Band 7. 2023a. https://www.mi.com/es/product/xiaomi-smart-band-7/
- [Background] Xiaomi. Xiaomi Smart Band 8. 2023b. https://www.mi.com/es/product/xiaomi-smart-band-8/
- [Background] Zarit SH, Anthony CR, Boutselis M. Interventions with care givers of dementia patients: comparison of two approaches. Psychol Aging. 1987 Sep;2(3):225-32. doi: 10.1037//0882-7974.2.3.225. PMID 3268213
- [Background] Zarit SH, Reever KE, Bach-Peterson J. Relatives of the impaired elderly: correlates of feelings of burden. Gerontologist. 1980 Dec;20(6):649-55. doi: 10.1093/geront/20.6.649. No abstract available. PMID 7203086
- [Result] Concheiro-Moscoso P, Groba B, Alvarez-Estevez D, Miranda-Duro MDC, Pousada T, Nieto-Riveiro L, Mejuto-Muino FJ, Pereira J. Quality of Sleep Data Validation From the Xiaomi Mi Band 5 Against Polysomnography: Comparison Study. J Med Internet Res. 2023 May 19;25:e42073. doi: 10.2196/42073. PMID 37204853